CLINICAL TRIAL: NCT00219882
Title: A Phase I Safety and Dose Finding Study of Orally Administered Curcuminoids in Adult Subjects With Cystic Fibrosis Who Are Homozygous for Delta F508 Cystic Fibrosis Transmembrane Conductance Regulator (ΔF508 CFTR) Mutation
Brief Title: Safety Study of Orally Administered Curcuminoids in Adult Subjects With Cystic Fibrosis
Acronym: SEER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ramsey, Bonnie, MD (Individual)
Collaborators: Seer Pharmaceuticals (Industry); CF Therapeutics Development Network Coordinating Center (Network); Cystic Fibrosis Foundation (Other)
Responsible Party: Chris Goss, MD, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEER-106
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2007-12-25 (Estimated); Status verified 2007-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; curcuminoids; turmeric root extract; nasal potential difference (NPD); sweat chloride
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): standardized turmeric root extract
  Interventions: Drug: standardized turmeric root extract

INTERVENTIONS:
Drug: standardized turmeric root extract — 1.5 gm of standardized tumeric root extract three times per day for seven consecutive days, followed by 3 gm of standardized tumeric root extract three times per day for seven consecutive days
  Other Names: AFI Curcuminoids

SUMMARY:
The purpose of this study is to assess the safety of advancing doses of curcuminoids administered orally for fourteen consecutive days in adult subjects with cystic fibrosis (CF) who are homozygous for ΔF508 CFTR.

DETAILED DESCRIPTION:
The drug substance being studied is curcumin. Curcumin (diferuloylmethane) is a major constituent in the spice turmeric, which is used as a food worldwide.

The pharmacologic rationale for studying curcumin for the treatment of cystic fibrosis is the potential for curcumin to help correct a deficiency of the cystic fibrosis transmembrane regulator (CFTR) protein. Cystic fibrosis results from a mutation of the CFTR gene, which produces abnormal CFTR protein that does properly transport chloride ion and water in the lung leading to abnormal mucus production. Curcumin is a potent inhibitor of the endoplasmic reticulum (ER) Ca2+ pump, and lowers ER calcium concentration. This may allow abnormal CFTR protein to function properly as a chloride channel and correct the cystic fibrosis defect. If this is successful, this effect could be measured as a decrease in the nasal potential difference (NPD) and sweat chloride in cystic fibrosis patients.

The primary objective of this study is to assess the safety of advancing doses of curcuminoids administered orally for fourteen consecutive days in adult subjects with cystic fibrosis (CF) who are homozygous for ΔF508 CFTR. The secondary objectives are to obtain pharmacokinetic data for oral curcumoniods in CF subjects and to assess the effectiveness of curcuminoids to alter nasal potential difference (NPD) and seat chloride concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 40 years of age.
* Documented history of being homozygous for ΔF508 CFTR genotype.
* Able to perform spirometry maneuvers, and have a forced expiratory volume at 1 second (FEV1) greater than or equal to 30% of predicted normal for age, gender, and height (Knudson standards) at screening.
* Oxygen saturation (as measured by pulse oximetry) > 90% on room air at screening.
* Clinically stable with no evidence of acute upper or lower respiratory tract infection.
* Non-smoker for at least 6 months prior to screening.
* Able to understand and sign a written informed consent and comply with the requirements of the study.

Exclusion Criteria:

* Diagnosis of acute pulmonary exacerbation (PE) requiring antibiotic intervention within 4 weeks prior to screening.
* Patient reported history of viral upper respiratory tract infection within 2 weeks prior to screening.
* History of major complications of lung disease (including recent massive hemoptysis or pneumothorax) within two months prior to screening Visit.
* Acute nosebleeds within 14 days prior to screening.
* Nasal surgery within 4 weeks prior to screening.
* Begun use of nasal antibiotics, nasal steroids, nasal cromolyn, nasal atrovent, nasal phenylephrine, or oxymetazoline within 14 days prior to screening.
* Chest x-ray at screening or within 3 months of screening with abnormalities suggesting clinically significant active pulmonary disease other than cystic fibrosis, and/or new CF-specific changes including atelectasis, small pneumothoraces, or pneumonia.
* EKG at screening which shows clinically significant abnormality including prolonged QTc, bundle branch block, rhythm other than sinus, evidence of ischemic heart disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2005-04; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 14 days of treatment with orally administered curcuminoids as assessed by adverse events, laboratory parameters, and spirometry. | 14 days

SECONDARY OUTCOMES:
(1) Pharmacokinetics of repeated doses of orally administered curcuminoids. (2) Change in nasal potential difference (NPD) measurements. (3) Change in sweat chloride measurements. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris Goss, MD, MSc, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Washington, Seattle, Washington